CLINICAL TRIAL: NCT00919828
Title: Adherent Monitoring of Congestive Heart Failure During Therapy for Excess Fluid Study
Brief Title: Monitor Patients With Acute Heart Failure
Acronym: ACUTE
Status: Completed | Type: Observational
Sponsor: Corventis, Inc. (Industry)
Responsible Party: Madhuri Bhat, VP Regulatory and Clinical affairs, Corventis
Other Study IDs: COR-2009-003
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Avivo System — Non invasive external monitoring device
  Other Names: external monitoring systems

SUMMARY:
This is a prospective, multi-center, non-randomized study to evaluate performance of an external monitor for heart failure patients

DETAILED DESCRIPTION:
External monitoring of heart failure patients with the AVIVO System.

ELIGIBILITY:
Inclusion Criteria:

* Is female or male, 18 years of age or older
* Has an ejection fraction of 40% reported within 12 months of enrollment
* Having acute decompensated heart failure and receiving treatment for fluid overload

Exclusion Criteria:

* Is participating in another clinical study that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)